CLINICAL TRIAL: NCT03499717
Title: Generalizability and Spread of an Evidenced-based Fall Prevention Toolkit: Fall TIPS (Tailoring Interventions for Patient Safety)
Brief Title: Generalizability and Spread of an Evidenced-based Fall Prevention Toolkit: Fall TIPS
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Montefiore Medical Center (Other); Partners HealthCare (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Patricia C. Dykes, Program Director, Center for Patient Safety Research and Practice, Brigham and Women's Hospital
Other Study IDs: 2017P000670
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Patient Fall
Keywords: Fall Risk; Patient Falls; Fall Prevention; Patient Safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of our project is to evaluate the effectiveness of the Fall TIPS program with regard to inpatient falls and fall-related injuries.

DETAILED DESCRIPTION:
This study will explore the effectiveness of the Fall TIPS (Tailoring Interventions for Patient Safety) program in regard to inpatient falls and fall-related injuries in three large hospital systems with different Electronic Medical Records (EMRs). We will collect and evaluate data on the perceived effectiveness of the Fall TIPS implementation process along with stakeholders' views of the toolkit. We will use an interrupted time series approach for evaluation of pre and post-Fall TIPS data related to patient falls and injurious falls. We will systematically analyze the costs and benefits of the Fall TIPS program from two perspectives: (1) the hospital, and (2) society as a whole. The hospital perspective will assist other hospitals in evaluating the decision to invest in implementing and adopting the Fall TIPS program, while the societal perspective will be instructive from a public policy stance

By the end of the study, we will produce a set of recommendations to facilitate adoption, implementation, and maintenance of the Fall TIPS program, along with a manuscript that will answer the following research questions:

1. Does Fall TIPS reduce the incidence of falls and injurious falls?
2. Were there differences in Fall TIPS effectiveness among different healthcare systems and hospitals as well as variations associated with differing patient characteristics (gender, age, ethnic/racial), EMRs, and degrees of adherence with the Fall TIPS protocol?
3. Do the benefits associated with Fall TIPS outweigh the costs from hospital and societal perspectives?
4. What Fall TIPS components were most/least useful and what recommendations will improve the overall utility and ease of use of the Fall TIPS Toolkit?
5. What aspects of the implementation model were most/least helpful for promoting Fall TIPS adoption and use?

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to medical, surgical, neurology and oncology units at participating hospitals during the time of the study

Exclusion Criteria:

* Anyone who does not meet the inclusion criteria

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all adult patients admitted to medical, surgical, neurology and oncology units at participating hospitals during the time of the study. Participating hospitals include the Partners Healthcare System, Montefiore Medical Center, and NewYork-Presbyterian/Columbia University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 37231 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Falls | 1/1/2014-12/31/2020
  Prevalence of patient falls in the study population

SECONDARY OUTCOMES:
Falls with Injury | 1/1/2014-12/31/2020
  Prevalence of patient falls with injury in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Dykes, MA,Ph.D,RN, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Result] Dykes PC, Burns Z, Adelman J, Benneyan J, Bogaisky M, Carter E, Ergai A, Lindros ME, Lipsitz SR, Scanlan M, Shaykevich S, Bates DW. Evaluation of a Patient-Centered Fall-Prevention Tool Kit to Reduce Falls and Injuries: A Nonrandomized Controlled Trial. JAMA Netw Open. 2020 Nov 2;3(11):e2025889. doi: 10.1001/jamanetworkopen.2020.25889. PMID 33201236
- See also: Evaluation of a Patient-Centered Fall-Prevention Tool Kit to Reduce Falls and Injuries: A Nonrandomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/33201236/